CLINICAL TRIAL: NCT04228601
Title: A Phase Ib/II Study to Assess the Tolerability, Safety and Efficacy of Fluzoparib in Combination With mFOLFIRINOX Followed by Fluzoparib Maintenance Monotherapy in Patients With Advanced Pancreatic Cancer
Brief Title: A Study of Fluzoparib in Combination With mFOLFIRINOX in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR3162-Ib/II-112
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluzoparib+mFOLFIRINOX (Experimental): Fluzoparib+mFOLFIRINOX followed by Fluzoparib maintenance monotherapy
  Interventions: Drug: Fluzoparib; Drug: mFOLFIRINOX
- Placebo+mFOLFIRINOX (Placebo Comparator): Placebo+mFOLFIRINOX followed by placebo maintenance monotherapy
  Interventions: Drug: Fluzoparib placebo; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Fluzoparib — PARP
  Other Names: SHR3162
  Arms: Fluzoparib+mFOLFIRINOX
Drug: Fluzoparib placebo — Placebo
  Arms: Placebo+mFOLFIRINOX
Drug: mFOLFIRINOX — mFOLFIRINOX

SUMMARY:
The study is being conducted to: a) evaluate the tolerability and safety of the co-administration of Fluzoparib and mFOLFIRINOX followed by Fluzoparib Maintenance Monotherapy in patients with advanced pancreatic cancer, and establish the maximum tolerated dose and recommended phase II dose of the combination; and b) assess the efficacy of the co-administration of Fluzoparib and mFOLFIRINOX followed by Fluzoparib Maintenance Monotherapy in patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Expected survival ≥ 6 months.
* Histologically or cytologically confirmed local advanced/metastatic pancreas adenocarcinoma.
* Documented mutation in germline BRCA1/2 or PALB2 that is predicted to be deleterious or suspected deleterious.
* Adequate organ performance based on laboratory blood tests.
* Presence of at least of one measurable lesion in agreement to RECIST criteria.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have received any chemotherapy for the treatment of pancreatic cancer prior to entering the study.
* Previous treatment with any poly ADP-ribose polymerase (PARP) inhibitor.
* Patients who have had radiotherapy or participated in another clinical trial with any investigational agents within 28 days of enrolment (Day 1 visit).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin, irinotecan, 5-Fluorouracil or other agents used in the study.
* Previous treatment using CYP3A4 inducers within 3 weeks or inhibitors within 2 weeks of enrolment (Day 1 visit).
* Patients with known or suspected brain metastasis.
* Significant cardiovascular disease such as New York Heart Associate Class III/IV, cardiac failure, myocardial infarction, unstable arrhythmia, or evidence of ischemia on ECG within 6 months prior to enrolment.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Patients with second primary cancer except curatively treated in-situ cancer or slowly progressing malignancy.
* Known active hepatitis B or C infection.
* History of immunodeficiency (including HIV infection) or organ transplantation.
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Phase Ib：Number of Participants With a Dose Limited Toxicity | Within 28 Days after The First Dose
  Number of Participants With a Dose Limited Toxicity
Phase Ib：Maximum Tolerated Dose | Up to 8 months
  Maximum Tolerated Dose
Phase Ib：Recommended Phase 2 Dose | Up to 2 years
  Recommended Phase 2 Dose
Phase II：Objective Response Rate | From Week 9 until documented disease progression or study discontinuation (approximately up to 24 months)
  Objective response rate according to RECIST 1.1

SECONDARY OUTCOMES:
Adverse events evaluated by NCI CTCAE v5.0 | From the first drug administration to within 30 days for the last drug dose
  Incidence of adverse events and associated dose of Fluzoparib
Disease Control Rate | From Week 9 until documented disease progression or study discontinuation (approximately up to 24 months)
  Disease control rate according to RECIST 1.1
Duration of Response | Up to 2 years
  Duration of Response
Progression-Free-Survival | Up to 2 years
  Time from randomisation until the date of objective radiological disease progression according to RECIST v1.1 or death
Overall-Survival | Up to 2 years
  Time from the date of randomization until death due to any cause
Area under the curve (AUC) | 1 year
  Area under the plasma concentration time curve from 0 to 24 hours for Fluroparib
Maximum concentration (Cmax) | 1 year
  Maximum observed plasma concentration for Fluzoparib
Time to maximum concentration (Tmax) | 1 year
  Time to maximum plasma concentration for Fluzoparib

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, M.D., Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wei M, Liu R, Xu Y, Chen X, Liu C, Bai X, Zhang X, Gao S, Li J, Sheng Z, Lian J, Wang W, Zhang J, Shi S, Xu J, Yu X. Phase 1b study of first-line fuzuloparib combined with modified FOLFIRINOX followed by fuzuloparib maintenance monotherapy in pancreatic adenocarcinoma. BMC Med. 2024 Sep 4;22(1):365. doi: 10.1186/s12916-024-03581-y. PMID 39232761